CLINICAL TRIAL: NCT01188213
Title: Efficacy of Methylsulfonylmethane Supplementation on Osteoarthritis of The Knee: A Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Other Study IDs: 13/05
Record Dates: First submitted 2010-08-21; First posted 2010-08-25 (Estimated); Last update posted 2010-08-25 (Estimated); Status verified 2005-05

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — dimethyl sulfone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Purified MSM (Experimental)
  Interventions: Dietary Supplement: Methylsulfonylmethane (MSM)

INTERVENTIONS:
Dietary Supplement: Methylsulfonylmethane (MSM)

SUMMARY:
The aim of this study was to determine the efficacy of methylsulfonylmethane (MSM) in treating patients with knee OA.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic knee OA for at least 6 months according to the clinical criteria of the American College of Rheumatology (ACR)
* radiographic confirmed knee OA according to the Kellgren & Lawrence scale

Exclusion Criteria:

* acute septic arthritis
* inflammatory arthritis
* any other type of arthritis
* history of knee buckling or recent knee injury
* lack of physical or mental bility to perform or comply with the treatment procedure
* diabetes mellitus
* fibromyalgia or other chronic pain syndromes
* concurrent anti-coagulant/anti-platelet drugs
* arthroscopy or intra-articular injections in the previous 3 months

Ages: 40 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
WOMAC questionnaire

REFERENCES:
- [Derived] Debbi EM, Agar G, Fichman G, Ziv YB, Kardosh R, Halperin N, Elbaz A, Beer Y, Debi R. Efficacy of methylsulfonylmethane supplementation on osteoarthritis of the knee: a randomized controlled study. BMC Complement Altern Med. 2011 Jun 27;11:50. doi: 10.1186/1472-6882-11-50. PMID 21708034